CLINICAL TRIAL: NCT02729194
Title: Pilot Study of Pazopanib With Low Fat Meal (PALM) in Advanced Renal Cell Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2016.013; HUM00111682 (Other: University of Michigan)
Record Dates: First submitted 2016-03-22; First posted 2016-04-06 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Registered subjects will take pazopanib by mouth with a low-fat meal (containing less than 400 calories and less than 10% fat or 10 grams per meal) approximately, some sample meals are described in appendix 1) every day in 14 day cycles, with a starting dose of 400 mg and adjusted for the next cycle (dose level +1:600 mg; dose level +2: 800 mg; dose level -1: 200 mg) based on toxicity assessment during or at the end of each cycle.
  Interventions: Drug: Pazopanib; Other: Low Fat Diet

INTERVENTIONS:
Drug: Pazopanib
Other: Low Fat Diet — Registered subjects will take pazopanib by mouth with a low-fat meal (containing less than 400 calories and less than 10% fat or 10 grams per meal.

SUMMARY:
Pazopanib is an orally administered multi-kinase inhibitor targeting VEGFR (vascular endothelial growth factor receptor), PDGFR (platelet derived growth factor) and c-kit, which are critical to growth and proliferation of neoplastic cells. Pazopanib has been FDA approved for advanced renal cell carcinoma (RCC) with a clear cell component. Conventional Pazopanib dosing WITHOUT FOOD is with an initial dose of 800 mg by mouth daily. Investigators hypothesize that administration of pazopanib with low fat meal would be safe and feasible with secondary implications of higher pazopanib levels; potentially translating into greater anti-tumor efficacy in advanced renal cell cancer, with significant cost savings. In the proposed pilot study, investigators seek to test the feasibility and practicality of this approach and gather preliminary data on adverse effects and the safety profile. Investigators hope to ameliorate any potential for greater toxicities with a dynamic dosing design that incorporates adverse events from each cycle into dosing for the next cycle and a structured symptom specific plan.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years of age) with unresectable locally advanced or metastatic renal cell carcinoma with a clear cell component.
* Subjects must have measurable disease per RECIST 1.1 criteria.
* Subjects must not have had prior pazopanib therapy.
* Subjects must have an ECOG (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.) performance status of less than or equal to 2.
* Up to 3 lines of prior VEGF (vascular endothelial growth factor) or VEGFR (vascular endothelial growth factor receptor) targeted therapy are permitted. Any prior therapy should have been completed ≥ 2 weeks prior to start of study therapy.
* Subjects may have received any number of the following therapies: cytokine therapy (e.g. high dose interleukin-2) or checkpoint inhibitor therapy (e.g. anti-PD1/PDL1, anti-CTLA4) or mTOR inhibitor therapy (e.g. everolimus, temsirolimus).
* Adequate organ and marrow function (Absolute neutrophil count > 1000/mm3, platelets > 100,000/mm3, aspartate aminotransferase/ alanine aminotransferase/ total bilirubin < 1.5 X ULN (upper limit of normal). Patients with Gilbert's disease are exempt.
* Subject must be willing and able to take pazopanib with a low-fat meal every day as specified in the protocol.
* Subjects must be willing and able to come off any PPI(proton pump inhibitor)/other strong CYP3A4 inhibitors or inducers/simvastatin.
* Ability to understand and the willingness to sign a written informed consent.
* All subjects, including those who are surgically sterilized, must be willing to use an effective method of contraception.

Exclusion Criteria:

* Any concurrent health condition that in the view of the treating physician would pose excessive risk to the patient if enrolled in the study.
* Subjects with a history of hemoptysis, cerebral hemorrhage, clinically significant GI hemorrhage, myocardial infarction within the past 6 months.
* Patients at significant risk for GI (gastrointestinal) perforation or fistula.
* Pregnant or nursing mothers.
* Untreated CNS (central nervous system) metastasis. If treated CNS metastasis/es, treatment of CNS disease (surgery or radiation) must have been completed at least 30 days prior to registration. Patients could still be on steroids.
* Subjects with known history of Cirrhosis, HIV, Hepatitis B or C.
* Averaged QTc baseline in 3 ECGs (electrocardiograms) at least 5 minutes apart of ≥450 ms.
* Congestive Heart Failure (NYHA Class III/IV) or LVEF (left ventricular ejection fraction) <50% at baseline.
* Uncontrolled hypertension (HTN) despite medical management (blood pressure (BP) ≥ 160/100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reimers MA, Shango MM, Daignault-Newton S, Dedinsky R, Karsies D, Kraft S, Riddle L, Felton JA, Wen B, Gersch C, Rae JM, Redman BG, Alva AS. Pazopanib with low fat meal (PALM) in advanced renal cell carcinoma. Invest New Drugs. 2019 Apr;37(2):323-330. doi: 10.1007/s10637-018-0692-8. Epub 2018 Nov 5. PMID 30393825

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib: Registered subjects will take pazopanib by mouth with a low-fat meal (containing less than 400 calories and less than 10% fat or 10 grams per meal) every day in 14 day cycles, with a starting dose of 400 mg and adjusted for the next cycle (dose level +1:600 mg; dose level +2: 800 mg; dose level -1: 200 mg) based on toxicity assessment during or at the end of each cycle.
Period: Overall Study
Arm/Group | Pazopanib
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Sixteen patients were enrolled in this study; three patients withdrew study consent prior to study completion.
Arm/Group | Pazopanib
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 60 [47 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Baseline Performance Status [Count of Participants; unit: Participants] — Baseline ECOG performance status. ECOG stands for Eastern Cooperative Oncology Group. The performance status is scale used by doctors and researchers to assess how the disease affects the daily living abilities of the patient.The scale ranges from 0 to 5 where 0 represents perfect health and 5 represents death.
  0=Fully active, able to carry on all pre-disease performance without restriction
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 11
    1 | 5
Histology [Count of Participants; unit: Participants] — Renal cell carcinoma cellular histology at baseline.
  Participants
    Pure Clear Cell | 11
    Mixed Histology | 5
Baseline Disease Site [Count of Participants; unit: Participants] — Sites of renal cell carcinoma metastasis at baseline.
  Participants
    Lung | 10
    Adrenal | 6
    Pancreas | 1
    Liver | 3
    Bone | 1
    Nephrectomy bed | 2
    Retroperitoneal and perisplenic nodule | 1
Heng Criteria Score [Count of Participants; unit: Participants] — The Heng Score for Metastatic Renal Cell Carcinoma (RCC) prognosis determines overall survival in patients treated with VEGF-targeted therapy using a scoring system that assigned points based off of a number of criteria.
  Score interpretation:
  0=Favorable 1-2=Intermediate
  ≥3=Poor
  Participants
    Favorable | 3
    Intermediate | 13
    Poor | 0
Number of Prior Therapies [Count of Participants; unit: Participants]
  No Prior Therapy | 12
  1 Prior Therapy | 3
  3 Prior Therapies | 1
Prior Therapy Type [Count of Participants; unit: Participants]
  Everolimus | 1
  High-dose IL-2 | 3
  Sunitinib | 1
  Nivolumab | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3 or 4 Adverse Events
Description: Number of grade 3 or 4 adverse events associated with pazopanib administered with a low fat meal by CTCAE version 4.0.
Time Frame: Through 12 weeks of treatment to 30 days post-treatment
Population: 16 participants were enrolled and treated.
Measure: Number; unit: adverse events
Arm/Group | Pazopanib
Number analyzed (Participants) | 16
adverse events
  Grade 3 adverse events associated with treatment | 5
  Grade 4 adverse events associated with treatment | 0

2. Primary Outcome: Number of Participants With Dose Reductions
Time Frame: 12 weeks
Population: 16 participants were enrolled. 13 of the 16 enrolled participants completed the 12 weeks of pazopanib therapy on study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
Participants | 3

3. Primary Outcome: Duration of Treatment
Description: The median duration of treatment will be reported.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: weeks
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
weeks | 12 [1 to 12]

4. Primary Outcome: Median Total Dose
Description: Median total dose given.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: mg
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
mg | 42,700 [1200 to 63,200]

5. Secondary Outcome: Percentage of Patients That Respond to Treatment (Overall Response) With Pazopanib Administered Along With a Low Fat Diet
Description: To estimate the overall response proportion to pazopanib administered with a low fat meal by RECIST 1.1 criteria. Overall response is defined as the number patients that experience Partial Response (PR) or Complete Response (CR).
  CR is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
  PR is defined as At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: 12 Weeks after start of study treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
percentage of participants | 38.46 [11 to 59]

6. Secondary Outcome: Number of Participants With Complete Response
Description: Complete response is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
Time Frame: 12 Weeks after start of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
Participants | 0

7. Secondary Outcome: Number of Patients With Partial Response
Description: Partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
Time Frame: 12 Weeks after start of study treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 13
Participants | 5

ADVERSE EVENTS:
Time Frame: Through 12 weeks of treatment up to 30 days post last treatment administration
Description: Adverse Events (AEs) were collected beginning at treatment start through 30 days post last treatment administration.
Arm/Group | Pazopanib
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=16)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=16)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 10 (12)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 8 (8)
Oral pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Pain (General disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (13)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 12 (15)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 5 (7)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 9 (10)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT02729194/Prot_SAP_000.pdf